CLINICAL TRIAL: NCT04570774
Title: Effect of Cerebral and Cerebellar Repetitive Transcranial Magnetic Stimulation on Motor Function in Stroke Patients
Brief Title: Effect of Cerebral and Cerebellar rTMS in Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-06-068
Record Dates: First submitted 2020-09-21; First posted 2020-09-30 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Repetitive Transcranial Magnetic Stimulation; rTMS; Motor Recovery
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facilitatory cerebral and cerebellar rTMS group (Experimental): Patients underwent 10 consecutive daily sessions of high-frequency repetitive transcranial magnetic stimulation (rTMS) over the affected primary motor cortex of the hand and high-frequency rTMS over the ipsilateral cerebellar hemisphere.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- Facilitatory cerebral rTMS group (Active Comparator): Patients underwent 10 consecutive daily sessions of high-frequency repetitive transcranial magnetic stimulation (rTMS) over the affected primary motor cortex of the hand and sham high-frequency rTMS over the ipsilateral cerebellar hemisphere.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- Inhibitory cerebral and cerebellar rTMS group (Experimental): Patients underwent 10 consecutive daily sessions of continous theta bust stimulation (cTBS) over the unaffected primary motor cortex of the hand and high-frequency rTMS over the ipsilateral cerebellar hemisphere.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation
- Inhibitory cerebral rTMS group (Active Comparator): Patients underwent 10 consecutive daily sessions of continous theta bust stimulation (cTBS) over the unaffected primary motor cortex of the hand and sham rTMS over the ipsilateral cerebellar hemisphere.
  Interventions: Procedure: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Repetitive transcranial magnetic stimulation — rTMS over cerebral motor cortex and cerebellar hemisphere

SUMMARY:
This study is based on the characteristics of motor learning theory and motor learning neural network to improve motor function in stroke patients. This study is to investigate whether the cerebral-cerebellar repetitive transcranial magnetic stimulation (rTMS) is effective in improving motor function compared to the conventional cerebral rTMS in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic stroke patients within 1 month after onset
* Moderate to severe motor impairment (Fugl-Meyer assessment <85)
* Cognitive and language functions to perform more than one step of command
* More than 19 years old

Exclusion Criteria:

* Contraindicated to rTMS
* Progressive or unstable stroke
* Pre-existing and active major neurological disease or major psychiatric disease
* A history of advanced liver, kidney, cardiac or pulmonary disease, a terminal medical diagnosis consistent with survival <1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Difference of upper limb motor score in Fugl-Meyer assessment | 2 weeks
  (upper limb motor score in Fugl-Meyer assessment at post-intervention) - (upper limb motor score in Fugl-Meyer assessment at baseline)
  Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available from the principal investigator upon reasonable request.